CLINICAL TRIAL: NCT06103344
Title: The Effect of 4-7-8 Breathing Exercise Training Given to Nursing Students on Sleep Quality: A Randomized-controlled Study
Brief Title: The Effect of 4-7-8 Breathing Exercise Training on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uğur Doğan (Other)
Responsible Party: Sponsor-Investigator, Uğur Doğan, Assistant Professor, Kilis 7 Aralik University
Organization: Kilis 7 Aralik University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kilis7AralikU-02
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Nursing Students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: 4-7-8 Breathing Exercise Training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: 4-7-8 Breathing Exercise Training — Participants in the intervention group will be taught 4-7-8 breathing exercises collectively, and the training will be repeated on specified days (twice a week for a total of 4 weeks). During the training, it will be checked whether each participant in the intervention group can perform the breathing exercise correctly and feedback will be given. Participants who fail to implement the exercise will be excluded from the study. 4-7-8 breathing exercise training, prepared in accordance with the literature, will be given by the assistant researcher who has training and certification in breathing exercises. Training will be planned in an empty classroom, for approximately 20 minutes and at the students' end time. Thus, educational activities in the institution will not be disrupted.
  Arms: Intervention

SUMMARY:
Research; it will be carried out Kilis 7 Aralik University Yusuf Serefoglu Health Sciences Faculty, Department of Nursing. The training will take approximately 20 minutes in an empty classroom and will be planned when the students' classes finish. Thus, educational activities in the institution will not be disrupted. Participants will be asked to do the taught exercise in half an hour before going to sleep every evening during the research period (4 weeks). Training will begin when the determined number of samples is reached. The training will be terminated when the 4-week research period determined to see the effect of the application expires.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* Studying in a nursing undergraduate program
* There is no condition that prevents nasal breathing (such as septal deviation)
* No known chronic sleeping disorder

Exclusion Criteria:

* No studying in a nursing undergraduate program
* There is condition that prevents nasal breathing (such as septal deviation)
* Having any chronic sleeping disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | This measurement will be repeated at the beginning of the study and at the end of the 4th week.
  Pittsburgh Sleep Quality Index evaluates sleep quality in the last month, contains a total of 24 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Doğan, PhD, Study Chair — Kilis 7 Aralik University
Locations (1):
- Kilis 7 Aralık University, Kilis, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No